CLINICAL TRIAL: NCT01478659
Title: The Effect of Fiber Snack Foods on Dietary Intake in Healthy Adults
Acronym: FIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: FIB
Record Dates: First submitted 2011-11-02; First posted 2011-11-23 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Fructooligosaccharide
Keywords: Diet; Fiber; Adult; Fructooligosaccharide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control bar and yogurt (Active Comparator)
  Interventions: Dietary Supplement: Control study food with no added fiber
- Fiber bar and yogurt (Experimental)
  Interventions: Dietary Supplement: Study food with added fiber

INTERVENTIONS:
Dietary Supplement: Control study food with no added fiber — Adults consuming their usual diet modified by incorporating yogurt and snack bars without added fiber.
  Arms: Control bar and yogurt
Dietary Supplement: Study food with added fiber — Adults consuming their usual diet modified by incorporating yogurt and snack bars containing 16 g of chicory root fiber (Frutalose®).
  Arms: Fiber bar and yogurt

SUMMARY:
The proposed study will be a randomized, double-blind, parallel-arm study. Participants will incorporate snack foods (bar/yogurt) containing 16 grams of fiber (fructooligosaccharide) or similar snack foods without the added fiber into their usual diets. The study period will include a 2-week pre-baseline assessment period and an 8-week treatment period. During the 2-week pre-baseline period no study foods will be consumed however dietary intake will be assessed using a 24-hour online diet recall program. The first week of the 8-week treatment will serve as an acclimation period where only one serving of the study foods will be given (8 grams of fiber) per day. Participants will receive two servings (16 grams of fiber) per day for weeks 2 through 8 of the treatment period and 24-hour online diet recalls will be completed during weeks 4, 6 and 8.

Hypothesis:

Adults aged 18 to 50 years consuming their usual diet modified by incorporating yogurt and snack bars containing 16 grams of chicory root fiber (Frutalose®) will decrease their usual dietary intake to a greater extent compared to participants who receive similar snack foods without the added fiber.

DETAILED DESCRIPTION:
The description of study activities is below:

Screening Period (approximately 2 weeks before randomization):

* Obtain height and weight
* Complete a 10-question survey about fruit, vegetable, and fiber intake
* Receive training on how to complete daily questionnaires online
* Complete the Global Physical Activity Questionnaire. This is a 16-question survey asking about physical activity in a typical week
* Complete the Eating Inventory. This is a 51-question survey that asks about your dietary habits and feelings related to food and eating
* Receive training on how to record your dietary intake using the ASA24. The ASA24 is a web-based interactive program that asks you to record the foods you ate during the previous day

Randomization:

* Measure weight, waist circumference, and body composition. We will use the BodPod to measure your body composition. The BodPod uses air displacement to measure body volume
* Receive dietary counseling on how to incorporate the study foods into your current diet. You will be asked to use these foods to replace foods you are currently eating
* Consume one study food per day for the first week and then 2 foods per day for weeks 2 through 8.
* Complete the 10-question online daily survey
* Complete 7 days of 24-hour dietary recalls using the ASA24 during weeks 4, 6, and 8

Final:

* Return any uneaten study foods.
* Measure weight, waist circumference, and body composition
* Complete the Global Physical Activity Questionnaire (GPAQ) and the Eating Inventory

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 50 years of age
* Internet access for the duration of the protocol
* BMI of 23.0 to < 30 kg/m2
* Usual fiber intake of <20 g/d based on FFQ such as the Block Fruit/Vegetable/Fiber Screener
* Weight stable (±5 lbs. last 3 months)
* Assessment of normal eating determined by the Eating Inventory
* Willing to eat yogurt and a granola-like snack bar daily for 8 weeks
* Willing to complete daily questionnaires and 28 dietary recalls over the 8 weeks
* Habitual breakfast consumer defined as eating breakfast (any food within 2 hours of waking) 5 or more days a week
* Willing to provide a social security number to receive study payment

Exclusion Criteria:

* Post-menopausal (self-reported no menstrual period for one year)
* Current smokers or tobacco users
* Based on Automated Self-Administered Diet History (ASA24) dietary intake data collected during pre-baseline period: Females eating less than 1200 kcal/day, males eating less than 1500 kcal/day or either or greater than 4000 kcal per day, consuming on average greater than 10 g dietary fiber/1000 kcal
* Unwilling to discontinue any prebiotic and fiber supplements, or probiotic supplement
* Antibiotic use within 2 months from study start
* Known food allergies
* Physician-diagnosed gastrointestinal disease or condition (such as ulcerative colitis, Crohn's disease, gastroparesis, cancer, peptic ulcer disease, Celiac disease, short bowel disease, ileostomy, colostomy other than GERD, constipation, diverticular disease)
* Taking prescribed medications other than oral contraceptives, seasonal allergy medications, cholesterol or blood pressure lowering medications, vitamins or minerals, baby aspirin
* Intake of >2 alcoholic drinks per day on average
* Purposeful exercise of >300 minutes per week on average
* Women who are lactating or know they are pregnant

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in pre-baseline and final average dietary intake | Pre-baseline Week and Week 8
  All participants will complete 24-hour online diet recalls during pre-baseline, week 4, 6 and 8 in order to determine if the addition of 16 g of fiber incorporated into snack bars and yogurt to the usual diets of mildly to moderately overweight adults results in reduced habitual energy intake compared to the addition of snack bars and yogurt without fiber.

SECONDARY OUTCOMES:
Change in anthropometrics from pre-baseline to week 8: height, weight, BMI, and body composition | Pre-baseline and final (week 8)
  All participants will have anthropometics measured at pre-baseline and again at the end of the study in order to determine if the addition of 16 g of fiber incorporated into snack bars and yogurt to the usual diets of mildly to moderately overweight adults results in reduced body weight and/or alter body composition compared to the addition of snack bars and yogurt without fiber.
Change in nutrient intakes from online diet recall program from pre-baseline to week 8 | Pre-baseline, Week 2, Week 4, and Week 8
  All participants will complete 24-hour online diet recalls during pre-baseline, week 4, week 6, and week 8 in order to determine if the addition of 16 g of fiber incorporated into snack bars and yogurt to the usual diets of mildly to moderately overweight adults alters macronutrient and micronutrients content within the diet compared to the addition of snack bars/yogurt without fiber.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Dahl, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States